CLINICAL TRIAL: NCT04700007
Title: Effect of Intradermal Morphine Application on Histaminergic and Non-histaminergic Itch and Related TRPV1 and Antihistamine Treatments (2nd Sub-project)
Brief Title: Evaluation of Peripheral Itch Mechanisms Following Injection of Morphine (Second Sub-Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20200084 2nd sub-project
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Capsaicin; Diphenhydramine; Histamine Antagonists; Morphine; Sodium Chloride; Histamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Drug: Capsaicin; Drug: Diphenhydramine; Drug: Morphine Chloride; Drug: Isotonic saline; Drug: Histamine

INTERVENTIONS:
Drug: Capsaicin — A capsaicin patch will be applied on a 3x3 cm squared area on the volar forearm. The patch will be left in place for 24h after which it will be removed.
Drug: Diphenhydramine — Diphenhydramin cream 1% (Restamine®) will be applied on a 3x3 cm squared predetermined area on the volar forearm for 24 hours.
  Other Names: Antihistamine
Drug: Morphine Chloride — Morphine solution (0.1mg/ml, Morphine Hydrochloride) 50 μl will be applied intradermally to the center of a predetermined area on the volar forearm by a 1 ml syringe.
Drug: Isotonic saline — injections of isotonic saline (0.05 ml, 0.9%) as vehicle will be performed.
Drug: Histamine — A small drop of histamine dihydrochloride (1%, in saline) will be applied to a previously determined area on the volar forearm followed by a prick through the drop.

SUMMARY:
The aim of our 2nd sub-project is to clarify if the capsaicin receptor TRPV1 is implicated in the mechanism of morphine-induced mast cell degranulation. Moreover, we also aim to clarify if the mechanism of opioid-induced itch relay on the histaminergic pathway by using the antihistamine (diphenhydramine) to suppress the release of histamine from peripheral mast cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Participants with any clinically significant abnormalities that in the opinion of the investigator may increase the risk associated with trial participation or may interfere with the interpretation of the trial results.
* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other addictive drugs
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics and pain killers as well as systemic or topical steroids.
* Participants with known allergy/discomfort to the opioid morphine and antihistamine.
* Skin diseases
* Moles, scars or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring itch intensity by computerized Visual Analog Scale Scoring | For 10 minutes
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring pain intensity by computerized Visual Analog Scale Scoring | For 10 minutes
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion measurement | After 15 minutes
  Superficial blood perfusion is measured by a Speckle contrast imager

SECONDARY OUTCOMES:
While size | After 15 minutes
  While size will be assessed using a ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Mech-Sense, Medicinsk Gastroenterologisk ambulatorium, Medicineshus, Aalborn Universitethospitalet, Aalborg, North Denmark, Denmark